CLINICAL TRIAL: NCT02332083
Title: Skilling-up Exercise for Elderly in Need of Care
Brief Title: Innovative Training Program for Elderly in Need of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Heiner Baur (PhD), PhD, Bern University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSc-study (Horgen)
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Poor Performance Status; Cognition - Other

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): T0 - intervention over 4 weeks with stochastic resonance whole-body vibration (SR-WBV) (start with 3 up to 6 Hz, noise 4) T1 - intervention 4 weeks (SR-WBV (start with 3 up to 6Hz, noise 4 & Exergame) - T2
  Interventions: Device: SR-WBV; Device: Exergame
- Sham Comparator (Sham Comparator): T0 - intervention 4 weeks (SR-WBV 1 Hz, noise 1) - T1 - intervention 4 weeks (SR-WBV 1 Hz, noise 1 & Aktiv Tramp) - T2
  Interventions: Other: SR-WBV; Device: Aktiv Tramp

INTERVENTIONS:
Device: SR-WBV — Participants will undergo a training program set over eight weeks, three times a week with 3 to 6 Hz, Noise 4.
  Other Names: SRT Zeptor® med
  Arms: Intervention group
Device: Exergame — Participants will undergo a training program set from week 5 to 8, three times a week over 20 minutes.
  Other Names: Virtual game board
  Arms: Intervention group
Other: SR-WBV — Participants will undergo a training program set over eight weeks three times a week with 1 Hz, Noise 1
  Other Names: SRT Zeptor® med
  Arms: Sham Comparator
Device: Aktiv Tramp — Participants will undergo a training program set from the 5 to 8 week, three times a week over 4 minutes.
  Other Names: Trampoline
  Arms: Sham Comparator

SUMMARY:
The goal of this randomized controlled study was to examine the effects of a 8 weeks innovative training regime (stochastic resonance whole-body vibration [SR-WBV] and virtual virtual games [VG]) in the skilling up phase on physical performance, cognition and falls in elderly in need of care population.

DETAILED DESCRIPTION:
Sensorimotor and strength exercise are methods to increase strength & power in the field of geriatrics. The question that arise what exercises are best suited to and most effective for elderly in need of care individuals. Such populations are advised first to enter a "skilling up program" before more traditional forms of training exercises are implemented.

Goals in the skilling up phase: improvement in neuromuscular control, postural control and strengthening of large muscle groups of the lower extremity.

The aim of the study in the skilling up phase:

Study the effect on physical performance Study the effects on muscle strength. Study the effects on cognition. The participants will be recruited in Canton Zurich, Swizerland and will be randomly allocated to an intervention group or sham group

ELIGIBILITY:
Inclusion Criteria:

* RAI (Resident Assessment Instrument) >0
* live in canton Zurich
* in terms of training load be resistant.

Exclusion Criteria:

* acut joint disease, acut thrombosis, acute fractures, acute infections, acute tissue damage, or acute

  * surgical scars
  * seniors with prosthesis.
  * alcoholic
  * acute joint disease, activated osteoarthritis, rheumatoid arthritis, acute lower limb
  * acute inflammation or infection tumors
  * fresh surgical wounds
  * severe migraine
  * epilepsy acute severe pain

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Short physical performance battery (SPBB) | 8 weeks
  The SPBB examines 3 areas of lower extremity function: standing balance (semi-tandem stand, side-by-side stand, full tandem stand), usual walking speed and ability to stand from a chair. These areas represent essential tasks important for independent living.

SECONDARY OUTCOMES:
Cognition | 8 weeks
  The trail-making test is a neuropsychological test of visual attention and task switching. The task requires a subject to 'connect-the-dots' of 25 consecutive targets on a sheet of paper. Two versions are available: A, in which the targets are all numbers (1,2,3, etc.), and B, in which the subject alternates between numbers and letters (1, A, 2, B, etc.). The goal of the subject is to finish the test as quickly as possible, and the time taken to complete the test is used as the primary performance metric.
The falls efficacy scale-international (FES-I) | 8 weeks
  The shortened version of the falls efficacy scale-international (FES-I): assess fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Baur, PD PhD, Principal Investigator — BUAS; Eling de Bruin, PD PhD, Study Chair — ETHZ
Locations (1):
- Bern University of Applied Science, Department Health, Bern, Switzerland